CLINICAL TRIAL: NCT06640101
Title: Effect of Inspiratory Muscle Training on Respiratory Function, Diaphragm Thickness, Balance Control, Exercise Capacity and Quality of Life in People After Stroke: a Randomized Controlled Trial
Brief Title: Effects of Inspiratory Muscle Training on Stroke Rehabilitation Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, LIU FANG, Principal Investigator, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: No.:HE-OT2023/13
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: Stroke; Inspiratory muscle training; Diaphragm; Balance control; Exercise capacity; Quality of life; Anticipatory postural adjustment time
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (sham IMT- stable group) (Sham Comparator): conventional treatment + sham IMT
  Interventions: Other: sham IMT; Other: Conventional treatment
- Group B (IMT-stable group) (Experimental): conventional treatment + target IMT while sitting on a stable surface
  Interventions: Other: IMT-stable group (sitting on a stable surface); Other: Conventional treatment
- Group C (IMT-unstable group) (Experimental): conventional treatment + target IMT while sitting on an unstable surface
  Interventions: Other: IMT-unstable group (sitting on an unstable surface); Other: Conventional treatment

INTERVENTIONS:
Other: sham IMT — with 10% maximum inspiratory pressure (MIP) as the training intensity, IMT will be conducted on a stable surface
  Arms: Group A (sham IMT- stable group)
Other: IMT-stable group (sitting on a stable surface) — 50% MIP as the training intensity, IMT will be conducted while sitting on a stable surface
  Arms: Group B (IMT-stable group)
Other: IMT-unstable group (sitting on an unstable surface) — 50% MIP as the training intensity, IMT will be conducted while sitting on an unstable surface
  Arms: Group C (IMT-unstable group)
Other: Conventional treatment — Participants in all groups will receive a standardised conventional rehabilitation protocol. It includes limb range of motion, muscle tone reduction, strengthening and endurance of limb muscles, transfer skills, task-directed movements, general gait training, and activities of daily living training.

SUMMARY:
This study is designed to explore the effects of a 4-week protocol of inspiratory muscle training (IMT) at 50% maximum inspiratory pressure (MIP) on respiratory function, diaphragm thickness, balance control, exercise capacity, and quality of life in people after stroke. To ascertain the effect of IMT on the relationship between diaphragm muscle contraction and activation of other trunk muscles, this study also explores whether any effect of the 4-week IMT protocol on balance control is associated with changes in the anticipatory posture adjustments (APAs) time - the onset time of postural muscles during a required task (e.g., the rapid shoulder flexion test).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years and < 80 years;
* breathing spontaneously;
* clinically diagnosed with ischemic and/or haemorrhagic stroke;
* duration of stroke from onset falls within 1 month to 12 months after diagnosis;
* no thoracic or abdominal surgery within the last 6 months;
* able to understand and follow verbal instructions;
* no facial palsy, or mild facial palsy without limitation of labial occlusion;
* able to maintain a resting sitting posture without feet support for at least 30 seconds;
* no cognitive impairment (Montreal Cognitive Assessment (MoCA) score ≥ 26);
* able to independently walk at least 10 meters with or without an assistive device.

Exclusion Criteria:

* acute myocardial infarction or acute heart failure;
* acute pain in any part of the body;
* with respiratory illness or positive clinical signs of impaired respiratory function (such as shortness of breath, hypoxemia, chronic cough and sputum retention);
* with chronic cardiovascular dysfunction;
* Trunk Impairment Scale (TIS) score ≥ 20.
* patient with a nasal feeding tube, tracheal tube and/or any condition that prevents the measurement or the implementation of the study procedure.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic thickness | baseline, after 4 weeks of intervention
  The diaphragmatic thickness of both the left and right diaphragms will be measured by ultrasound. (Mindray M9, Shenzhen, China).

SECONDARY OUTCOMES:
Maximum Inspiratory Pressure (MIP) | baseline, after 4 weeks of intervention
  Maximum Inspiratory Pressure (MIP) is a measure used in pulmonary function testing to assess the strength of the respiratory muscles, particularly the muscles used for inhalation. It will be measured using the spirometer.
Forced Vital Capacity (FVC) | baseline, after 4 weeks of intervention
  Forced Vital Capacity (FVC) is a measurement used in pulmonary function tests to assess lung function. It refers to the total volume of air that a person can forcibly exhale from their lungs after taking the deepest breath possible. It will be measured using the spirometer.
Forced Expiratory Volume in one second (FEV1) | baseline, after 4 weeks of intervention
  Forced Expiratory Volume in one second (FEV1) measures the volume of air a person can forcibly exhale in the first second of a forced breath. It will be measured using the spirometer.
Sitting Balance | baseline, after 4 weeks of intervention
  A force plate will be used to measure changes in the center of pressure during the performance of various tasks in sitting positions.
Trunk Impairment Scale (TIS) | baseline, after 4 weeks of intervention, 12-week follow-up after the end of intervention
  The TIS is a rating scale used to measure static sitting balance, dynamic sitting balance, and trunk coordination. The total TIS score ranges from 0 to 23 points, with a higher score indicating better trunk function.
Timed Up and Go Test (TUG) | baseline, after 4 weeks of intervention, 12-week follow-up after the end of intervention
  TUG is a test to measure the time that a participant needs to stand up from a standard armchair, walk a short distance of about 3 meters, turn around, walk back to the chair, and sit down again.
Falls efficacy scale international | baseline, after 4 weeks of intervention, 12-week follow-up after the end of intervention
  The Falls Efficacy Scale-International (FES-I) is a questionnaire measuring fear of falling in older adults. It has 16 items, scored from 1 to 4, with higher scores indicating greater fear. It's used in clinical settings to assess fall risk and tailor interventions.
6-Minute Walk Test | baseline, after 4 weeks of intervention
  The 6-Minute Walk Test (6MWT) measures how far someone can walk in six minutes. It assesses exercise capacity and mobility.
Stroke Impact Scale | baseline, after 4 weeks of intervention, 12-week follow-up after the end of intervention
  The Chinese version of the Stroke Impact Scale 3.0 (SIS) will be used to measure the quality of life. A higher overall score suggests better physical, emotional, and social functioning, while a lower score may indicate more significant impairment or limitations.
Trunk muscle activity | baseline, after 4 weeks of intervention
  Surface electromyography (sEMG) (Noraxon USA, Inc., Scottsdale, AZ, USA) will be used to measure the bilateral muscle activity of the erector spinae, rectus abdominis, external oblique muscle, internal oblique muscle, and transversus abdominis during sitting balance tests on the force plate.
Anticipatory posture adjustments (APAs) time of trunk muscles | baseline, after 4 weeks of intervention
  Participants will be requested to perform a rapid shoulder flexion test on the force plate. Surface electromyography (sEMG) (Noraxon USA, Inc., Scottsdale, AZ, USA) will be used to measure Anticipatory posture adjustments (APAs) time of trunk muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, None Selected, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu F, Jones AY, Tsang RC, Yam TT, Tsang WW. Inspiratory muscle training with balance challenge improves diaphragmatic thickness, respiratory function, balance, exercise capacity and quality of life in people after stroke: a randomised trial. J Physiother. 2026 Jan;72(1):42-52. doi: 10.1016/j.jphys.2025.12.004. Epub 2025 Dec 20. PMID 41423385

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT06640101/Prot_SAP_002.pdf
  • Informed Consent Form (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT06640101/ICF_003.pdf